CLINICAL TRIAL: NCT06072300
Title: The Effects of Physical Activity Calorie Equivalent (PACE) Labelling on Hot Beverage Transactions From Vending Machines: Stepped-wedge Cluster Randomised Trial
Brief Title: Effects of Physical Activity Calorie Equivalent Labelling on Hot Drink Vending Transactions
Acronym: PACE-VEND
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Amanda Daley, Professor, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1307
Record Dates: First submitted 2023-09-29; First posted 2023-10-10 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Averaged Kilocalories Per Beverage Transaction; Proportion of Total High Calorie Beverages; Total Number of Beverage Transactions

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomised trial
Masking Description: No individuals other than the University facility staff assisting with this study will be aware of the aims of the research. It is not possible to blind the trial statistician to the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The placement of physical activity calorie equivalent labelling on beverage vending machines
  Interventions: Behavioral: Physical activity calorie equivalent labelling
- Comparator (No Intervention): No physical activity calorie equivalent labelling on beverage vending machines

INTERVENTIONS:
Behavioral: Physical activity calorie equivalent labelling — Physical activity calorie equivalent labelling on beverage vending machines
  Other Names: PACE labelling
  Arms: Intervention

SUMMARY:
Food nutritional labels are one way to support people to make more informed, healthier food choices. However, there is limited evidence from trials showing that nutrition information on food or drinks is changing the food purchasing or food/beverage consumption behaviours. Many people do not understand the meaning of kilocalories (kcals, calories) or grams of fat displayed on food labels, and often underestimate the number of calories when labelling is not provided. An alternative or complementary approach to current nutrition labelling, is to provide calorie information with a clear interpretation of what the calorie content of the food item/meal or beverage means in terms of energy expenditure. This approach has been called physical activity calorie equivalent (or expenditure) labelling (PACE), which aims to show the public how many minutes (or miles/kilometres) of physical activity (e.g. walking or running) are equivalent to the calories contained in food/beverages. For example, "the calories in this chocolate bar require 95 minutes of walking to burn off". One context in which the public consume a lot of calories is from vending machines. We hypothesise that providing consumers with PACE information on hot beverage vending machines will reduce the average number of calories per transaction dispensed from the vending machines compared with when no PACE information/labelling is presented on vending machines. The study will adopt what is called a stepped wedge randomised controlled trial design involving 42 hot beverage vending machines in 27 buildings (clusters). Clusters will be randomly allocated to one of eight sequences across 24 weeks, which will dictate the time (weeks) at which clusters display the vending machine PACE labelling intervention. Weeks one to four will constitute a baseline period, during which the data will be collected from all vending machines without PACE labelling in place. This will be followed by 20 weeks during which the PACE labelling intervention will be introduced and maintained at each building according to a stepped wedge design (Figure 2). Specifically, every two weeks, three or four clusters will move to the intervention condition. The number of transactions from the vending machines will be collected over the study period and we will compare the number of transactions in the weeks when the PACE labelling is displayed compared to when it was not.

DETAILED DESCRIPTION:
The study will adopt a stepped wedge randomised controlled trial (SW-CRT) design involving 42 hot beverage vending machines in 27 buildings (clusters). Clusters will be randomly allocated to one of eight sequences across 24 weeks, which will dictate the time at which clusters implement the vending machine PACE labelling intervention (condition). Weeks one to four will constitute a baseline period, during which the data will be collected from all vending machines without PACE labelling in place. This will be followed by 20 weeks during which the PACE labelling intervention will be introduced and maintained at each building according to the SW-CRT design. Specifically, every two weeks, three clusters will move from no PACE labelling to the intervention condition.

All vending machines have the same seven hot beverage options (hot water, espresso, black coffee, flat white coffee, cappuccino, mocha, latte macchiato and hot chocolate). When vending machines are randomised to display the PACE labelling, they will display sticker labels showing the number of calories and minutes walking (averaged speed) to expend the calories of each beverage.

Data for the number and type of hot beverages transactions will be collected every week or two weeks from each vending machine. Photograph date stamped evidence of the number of transactions beverages will be collected.

The primary outcome will be averaged kilocalories (kcals) per transaction. We will evaluate the proportion of total drinks dispensed that are high calorie, and so each beverage dispensed will be dichotomised as being high-calorie or not high-calorie. It is possible people choose not to have a beverage at all in response to the intervention. A secondary aim is to compare total number of transactions of beverages between the PACE labelling and comparator condition.

Randomisation will be performed at the cluster (building) level. A total of 27 buildings will be randomised to one of eight sequence using covariate constrained randomisation (CCR) to ensure a balance of several cluster-level covariates. The covariates included in this constrained randomisation procedure will be: type of building, number of vending machines in each building/cluster and average baseline (weeks 1-4) mocha transactions per cluster (most caloric beverage) (defined as low, medium and high). Three days prior to the next batch of clusters transitioning to the intervention condition, the trial statistician will reveal the subsequent vending machines that have been randomised to display the PACE labelling in line with the study plan. The allocation sequence will not be known to researchers except for the trial statisticians.

ELIGIBILITY:
Inclusion Criteria:

All vending machines within a cluster need to be self-service customer operated.

Vending machines need to be operated and maintained by the participating University

All vending machines within a cluster need to dispense the same hot beverages of interest

All vending machines in the cluster electronically record transactions of the hot beverages.

Exclusion Criteria:

Vending machines or clusters not meeting the inclusion criteria

Not able to access the vending machine for the purpose of this study

Any vending machine the ethics committee feel it is inappropriate to collect data from (e.g. near a medical facility), in which the case the whole cluster (location) will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Averaged kilocalories (kcals) per transaction | six months
  Averaged kilocalories (kcals) per transaction

SECONDARY OUTCOMES:
Total drinks dispensed that are high calorie | Six months
  Total drinks dispensed that are high calorie
Total number of transactions of beverages | Six months
  Total number of transactions of beverages

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Daley, PhD, Principal Investigator — Loughborough University
Locations (1):
- School of Sport, Exercise and Health Sciences, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We plan to make available the study data in the University data depository once it is completed and published.
Supporting Information: CSR
Time Frame: Data will be available after the study is completed and published
Access Criteria: On request from the contacts listed